CLINICAL TRIAL: NCT02274831
Title: You Have Got Got Mail....and Need Follow Up
Brief Title: EMail Reminder to Follow up With Primary Physician
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Trinity Health Michigan (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: StJosephMHS
Record Dates: First submitted 2014-10-23; First posted 2014-10-24 (Estimated); Last update posted 2014-10-24 (Estimated); Status verified 2014-10

CONDITIONS: Act Code - Emergency

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Email Group (Experimental): Includes receiving standard of care discharge instructions plus an email after being discharged home from the emergency department, reinforcing their discharge instructions. Included in the email is their physician's name and recommended timing of follow-up visit.
  Interventions: Other: Email Reminder of need to follow up with primary physician
- Standard of Care (No Intervention): Includes standard of care discharge instructions after being discharged from the emergency department. This included receiving paper copies of their discharge instructions.

INTERVENTIONS:
Other: Email Reminder of need to follow up with primary physician
  Arms: Email Group

SUMMARY:
The purpose of this study is to see if patients who receive an email reinforcing their discharge instructions after being discharged from the emergency department will have an affect on follow-up care with their primary physician.

DETAILED DESCRIPTION:
When a patient is treated in the emergency department (ED), they experience a whirlwind of care involving multiple diagnostics and treatments. They are often discharged home with instructions to follow up with their primary care physician. This follow up care is crucial to ensuring optimal patient outcomes and re-establishing continuity of care. Despite efforts to communicate clearly and effectively, ED patients often have difficulty understanding their follow-up care instructions. Several different methods have been employed to attempt to improve the follow-up rates after emergency department care, including providing patients with an easily read, printed copy of discharge instructions, having a nurse or mid-level provider call patients days after discharge from the ED to ensure that they understood discharge instructions. One medium for communication that has become increasingly relevant in recent years is electronic mail (email). Because of its pervasiveness and relative ease of use, email offers a potentially valuable resource for augmenting and improving communication between physicians and patients. This study will assess whether an email reminder with follow up instructions one day after ED visit occurs will increase follow up rates and timely follow up rates.

ELIGIBILITY:
Inclusion Criteria:

* 1. Patients triaged to category 2, 3, and 4 and placed in a room for care at St. Joseph Mercy Hospital-Ann Arbor Emergency Department 2. Primarily English speaking. 3. >18 years of age 4. Have a primary physician who is part of Integrated Health Associates 5. Have access to an email account

Exclusion Criteria:

* 1. Patients triaged to category 1 or 5 placed in a room at Stl Joseph Mercy Hospital-Ann Arbor (category 1 patients are not typically discharged home from the hospital. Category 5 patients could potentially be interfered with if attempting implementation of the communication instrument. Category 5 patients are typically very straightforward visits with minimal requirement for follow-up appointments) 2. Patients < age 18 3. Prisoners or institutionalized persons 4. Patients with a mental-health related chief complaint 5. Not primarily English speaking (the potential language barriers could interfere with ability to communicate via email which will be written in English) 6. Under temporary or permanent custodianship (used as a surrogate for ongoing lack of mental competence or consciousness) 7. Prior participation in this study. (A patient may only participate once).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 577 (Actual)
Dates: Start 2011-08; Primary Completion 2014-03 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
Successful follow-up with primary care physician | 10 days
  Review of medical records at primary care physician's office by one of two physician investigators